CLINICAL TRIAL: NCT01289470
Title: Clinical Assessment of Nonin 7600 Near Infrared Spectroscopy (NIRS) Tissue Oximetry During Cardiovascular Surgery
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP1881
Record Dates: First submitted 2011-01-14; First posted 2011-02-03 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery
Keywords: NIRS Technology; Cardiovascular surgery; valvular surgery with cardiopulmonary bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An observational study designed to evaluate the performance of a new Near Infrared Spectroscopy (NIRS) tissue oximeter device in the clinical setting, including a cerebral sensor and peripheral sensor. Fifty patients who are undergoing open-heart surgery will be enrolled and tissue oximetry measurement will be collected throughout the surgical procedure and for up to 24 hours following surgery. Tissue oximeter measurement of the brain and skeletal tissue will be added to the standard intra-operative patient monitoring. Measures of delirium will be collected using a standardized questionnaire. The relationship between cerebral oximetry measures and delirium scores will be explored.

DETAILED DESCRIPTION:
See Eligibility Criteria section

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Weigh at least 40 kg
* Undergoing Coronary Artery Bypass Graft (CABG) and/or valvular surgery requiring the use of Cardio Pulmonary Bypass (CPB) or Left Ventricular Assist Device (LVAD), inclusive of any concomitant procedure
* Willing and able to provide informed consent
* Able to communicate and read in English

Exclusion Criteria:

* Emergency procedure such that informed consent may not be obtained
* Known cognitive impairment, history of delirium or dementia
* Known hemodialysis or fistula graft
* Delirium Observation Score (DOS) Score of >6 prior to surgery
* Pre-existing skin condition at the site of sensor application (e.g. eczema, dermatitis)
* Any known contraindication or sensitivity to the cerebral oximeter sensor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Coronary Artery Bypass Graft (CABG) and valvular surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Percent of time Regional Oxygen Saturation (rSO2) values are registered during open heart surgery. | Completion of cardiovascular surgery

SECONDARY OUTCOMES:
Correlation between delirium outcome scale and Regional Oxygen Saturation (rSO2) values. | Patient discharge (on average 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Solomon Aronson, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States